CLINICAL TRIAL: NCT03742388
Title: A Genomic Analysis on the Evolution of Epithelia Ovarian Tumors
Brief Title: A Genomic Analysis of Evolution of Epithelia Ovarian Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-BORDERLINE
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Epithelial Ovarian Cancer; Epithelial Ovarian Tumor of Borderline Malignancy; Driving Mutations; Progression-free Survival
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissues for genomic analysis will be collected from paraffin section by microdissection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epithelial ovarian carcinomatous and borderline components sometimes appeared in one patient. This study aims to analyze the genomic patterns of the carcinomatous and borderline components in the ovarian epithelial tissues. These tissues will be collected from paraffin section by microdissection to distinguish normal, carcinomatous and borderline tissues.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary epithelial ovarian borderline tumor with cancer
* Signed an approved informed consents
* Feasible for sampling

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with diagnosis of primary epithelial ovarian borderline tumor with cancer will be included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-12-23 (Estimated); Study Completion 2020-12-23 (Estimated)

PRIMARY OUTCOMES:
Frequencies of somatic driving mutations | Two years
  The differences of frequencies of somatic driving mutations will be compared between normal, carcinomatous and borderline tissues.

SECONDARY OUTCOMES:
Progression-free survival | Five years
  Progression-free survival between patients with differential expressed multi-omics will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China